CLINICAL TRIAL: NCT06796296
Title: The Safety and Efficacy of Transanal Irrigation in Patients from Low Anterior Resection Syndrome After Rectal Cancer Surgery : a Multicenter Prospective Randomized Controlled Trial (TraLARS Study)
Brief Title: Transanal Irrigation for Low Anterior Resection Syndrome
Acronym: TraLARS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); National Cancer Center, Korea (Other Government); Seoul National University Boramae Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-2310-121-1479
Record Dates: First submitted 2024-12-13; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-11

CONDITIONS: Low Anterior Resection Syndrome; Rectal Cancer Surgery; Insomnia
Keywords: Transanal irrigation; Low anterior resection syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loperamide group (No Intervention): The group only takes loperamide in the evening (2mg once daily orally)
- Loperamide + Transanal irrigation (Experimental): The group takes Loperamide daily and undergoes transanal irrigation once or twice a week
  Interventions: Procedure: Transanal Irrigation (TAI)

INTERVENTIONS:
Procedure: Transanal Irrigation (TAI) — The combination of transanal irrigation (TAI) and Loperamide involves administering Loperamide orally, with a daily dosage of 2mg. This is complemented by the use of TAI, a method in which patients self-administer water into the rectum through an enema, aiming to enhance bowel management and potentially alleviate sysmptoms associated with LARS
  Arms: Loperamide + Transanal irrigation

SUMMARY:
The preservation surgery of the anal sphincter muscle has become the standard procedure in the treatment of rectal cancer and, thanks to advancements in surgical techniques, can now be performed for tumors located closer to the anus. This method allows patients to avoid a permanent artificial anus, maintaining continuity of the intestines and enabling bowel movements through the anus, making it a highly preferred procedure. Furthermore, advancements in various tumor treatments have led to improved long-term survival rates.

Preservation surgery of the anal sphincter muscle is commonly used in the treatment of rectal cancer, resulting in approximately 90% of patients experiencing changes in bowel habits after surgery. These changes include characteristic diarrhea, urgent bowel movements, frequent bowel movements, and fecal incontinence, collectively known as Anterior Resection Syndrome (ARS). Particularly in the case of low rectal cancer, it often manifests as Low Anterior Resection Syndrome (LARS). These symptoms are most severe immediately after surgery, generally persisting in a significant degree for 1-2 years, with some improvement over time. However, for many patients, LARS remains a lifelong challenge, significantly impacting their quality of life. Nighttime symptoms of LARS, in particular, have a profound effect on sleep quality, potentially leading to a decline in overall quality of life.

Currently, there is no definitive method to completely cure LARS, and the available approaches focus on empirical treatments or short-term symptom control using medications such as loperamide.

Loperamide directly affects the neuromuscular system of the intestine, reducing its motility. This prolongs the time food stays in the intestine, allowing sufficient absorption of moisture and electrolytes, consequently reducing symptoms of diarrhea. Loperamide is available in two forms: loperamide oxide and loperamide hydrochloride. While loperamide oxide products like Arestal® were prescribed by doctors until August 2017, the approval was revoked, leaving loperamide hydrochloride as the only form used domestically. It comes in a single product containing 2 mg of loperamide hydrochloride and a combination product with 0.25 mg of loperamide hydrochloride, a sterilizing agent in the intestine (e.g., acrylonitrile, berberine), and an antispasmodic.

Transanal irrigation (TAI) is a method where patients self-administer water into the rectum through an enema, physically cleansing the anus and rectum. This technique is often used for patients with chronic constipation or fecal incontinence. TAI has proven beneficial, particularly in improving symptoms for patients experiencing bowel dysfunction following sphincter-preserving surgery, especially for those who underwent low anterior resection.

However, there is currently no research on the utility and safety of TAI for LARS patients, specifically addressing whether it can improve the nighttime symptoms associated with LARS syndrome and enhance sleep quality. Therefore, this study aims to investigate the impact of TAI on the symptoms of LARS syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years and above.
* Patients who have undergone low or ultra-low anterior resection surgery for rectal cancer (within 15cm from the anal verge).
* Patients at least 24 months post-surgery without stoma.
* Patients evaluated with a major LARS score.
* Patients who comprehend and have the ability to participate in this clinical trial.

Exclusion Criteria:

* Patients with recurrent colorectal cancer.
* Patients with concomitant metastatic colorectal cancer.
* Patients requiring permanent colostomy.
* Patients who have undergone postoperative cancer radiation therapy.
* Patients with underlying conditions not controlled by internal medical treatment.
* Patients with inflammatory bowel disease (IBD).
* Patients with symptoms of constipation or diarrhea not controlled by medication.
* Patients with preoperative symptoms of fecal incontinence.
* Patients allergic to the investigational drug.
* Patients deemed unsuitable for clinical trial participation by the principal investigator and study personnel.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of major LARS | 4 weeks
  Patients are requested to answer the LARS score questionnaires at inclusion (0 week) and 4 weeks after intervention at the outpatient clinic.
  The score ranges from 0 to 42, with 0-20 signifying no LARS, 21-29 signifying minor LARS, and 30-42 signifying major LARS.
  Only patients with major LARS at 0 week are enrolled. Re-measure the LARS score at week 4 to see the rate of improvement (minor LARS or no LARS) in major LARS in both groups.

SECONDARY OUTCOMES:
The LARS (Low Anterior Resection Syndrome) score | 4 weeks
  A survey is conducted, scoring patient's symptoms related to LARS. It includes the LARS score with night-time symptoms.
Insomnia Severity Index score in Korean Validation | 4 weeks
  A survey is conducted, scoring patient's symptoms related to Insomnia.
European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | 4 weeks
  A survey is conducted, scoring patient's symptoms related to LARS and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongro-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided